CLINICAL TRIAL: NCT07168278
Title: Tenecteplase vs Medical Management in 4.5-24h Anterior Circulation Large Vessel Occlusion With no Access to EVT
Brief Title: Tenecteplase vs Medical Management in 4.5-24h LVO no Access to EVT
Acronym: TNK LATE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KY348
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion; Tenecteplase; Thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK (Experimental): Participants will receive intravenous tenecteplase at a dose of 0.25 mg/kg (max 25 mg) administered as a bolus after enrollment. Subsequent treatment will be administered with antiplatelet drugs, anticoagulation or combinations of these treatment modality according to national and institutional guidelines.
  Interventions: Drug: TNK
- Standard medical management (Placebo Comparator): Participants will receive antiplatelet drugs, anticoagulation or combinations of these treatment modality according to national and institutional guidelines.
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Drug: TNK — a dose of 0.25 mg/kg (max 25 mg) administered as a bolus
  Other Names: tenecteplase
  Arms: TNK
Drug: Standard medical treatment — antiplatelet drugs, anticoagulation or combinations of these treatment modality according to national and institutional guidelines.
  Other Names: standard treatment
  Arms: Standard medical management

SUMMARY:
The goal of this clinical trial is to learn if tenectplase works to acute ischemic stroke (AIS) with onset 4.5-9 hours. It will also learn about the safety of tenectplase in AIS with onset 4.5-9 hours. The main question it aims to answer is: Does tenectplase improve the 90-days functional outcome in participants with acute large vessel occlusion? Researchers will compare tenectplase thrombolysis to non-use to see if tenectplase works to improve the functional outcome in participants with onset 4.5-9 hours. Participants will:* Receive 0.25mg/kg (max 25mg) tenectplase at admission (after randomization) .* Receive neurological assessment at admission, Day 5-7 or on hospital discharge (whichever earlier). Audio or video of the assessment may be recorded if possible.* Receive brain CT + CT angiogram + CT perfusion and MRI after randomization, where the CT scan may be repetitive.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Acute ischemic stroke presenting in the 4.5 to 24 hour window from last seen well (including wake-up stroke and no witness stroke).
* Prestroke mRS 0-2
* NIHSS 6 to 25
* Aspect ≥ 7
* ICA terminus, M1, dominant M2 occlusion on CTA or MRA
* Clinical-imaging mismatch assessed by investigator
* Patients with no access to EVT at the time of randomization

Exclusion Criteria:

* Current or past history of significant bleeding over the past 6 months;
* History of intracranial hemorrhage (including possible subarachnoid hemorrhage or subarachnoid hemorrhage due to an aneurysm) or evidence or suspected intracranial hemorrhage;
* Known bleeding tendency;
* Recent severe or dangerous bleeding, or active ulcerative gastrointestinal disease;
* History of central nervous system injury (e.g., intracranial tumor, aneurysm, or arteriovenous malformation, intracranial or spinal surgery), or recent head injury；
* Tumors that increase risk of bleeding;
* Severe liver dysfunction, including liver failure, cirrhosis, portal hypertension (esophageal varices), and active hepatitis;
* Know arterial / venous malformation or aneurysm;
* Bacterial endocarditis, pericarditis, or acute pancreatitis;
* Patients receiving effective anticoagulant therapy (vitamin K antagonists with INR > 1.3, or other oral anticoagulants exceeding the upper limit of the corresponding standard range);
* Heparin use within the past 48 hours and prothrombin time exceeding the upper limit of the standard range;
* Over the past 3 months, undergone major surgery, organ biopsy, or suffered a serious injury;
* Over the past 2 weeks, receiving prolonged ( >2 minutes) cardiopulmonary resuscitation, childbirth, or non-stressful vascular puncture (such as subclavian or jugular vein puncture);
* Stroke episode occurred with epileptic seizure;
* History of stroke comorbid with diabetes;
* History of stroke over the past 3 months；
* Acute bleeding tendency, including platelet count below 100×10⁹/L or other conditions;
* SBP >185 mmHg or DBP >110 mmHg, or requiring intensive treatment (intravenous antihypertensive drugs) to lower blood pressure to within limits;
* Blood glucose <2.8 mmol/L or >22.2 mmol/L (<50 mg/dL or >400 mg/dL)；
* Patient life expectancy of less than 1 year;
* Simultaneous occlusion of multiple blood vessels, defined as bilateral MCAs or MCAs combined with the basilar artery;
* Pregnant women or nursing mothers；
* Patients with a low likelihood of 3-month follow-up；
* Over the past 3 months participated in other interventional clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with functional independence outcome (mRS 0-2) at day 90 | 90 days after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
The ordinal shift of modified Rankin Scale | 90 days after procedure
  The Modified Rankin Scale (mRS) measures degree of disability/dependence after a stroke, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death
Proportion of patients with functional independence outcome (mRS 0-1) at day 90 | 90 days after procedure
  Modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Recanalization of occlusion site according to the arterial occlusive lesion (AOL) scale | 24 hours after randomization
  It specifically measures the mechanical success of recanalization at the site of the original occlusion.The scale ranges from 0 to 3, with higher scores indicating better recanalization. Grade 0: No recanalization (persistent occlusion). Grade 1: Incomplete recanalization (partial reopening with minimal flow). Grade 2: Partial recanalization (significant flow but residual stenosis or thrombus). Grade 3: Complete recanalization (full restoration of flow with no residual occlusion).
Change in Neurological Function of Participants Assessed by National Institute of Health Stroke Scale | Baseline and 7-days after randomization (or at discharge)
  Zero indicates no stroke symptoms, 1-4 , 5-15, 16-20, 21-42 indicate minor, moderate, moderate to severe, and severe stroke, respectively.
Symptomatic intracranial hemorrhage (SICH) as defined by the Heidelberg Bleeding Classification | within 36 hours after randomization
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 24 hours , or any hemorrhage leading to death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No